CLINICAL TRIAL: NCT06706245
Title: Developing a Virtual Reality Training Tool for Exposure Therapy: Simulated Exposure Trainer (SET)
Acronym: SET-VR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bradley Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Joshua Kemp, Staff Clinician / Assistant Professor (Research), Bradley Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 841660; 1R41MH131229-01 (NIH); 5R41MH131229-02 (NIH)
Record Dates: First submitted 2024-11-19; First posted 2024-11-26 (Actual); Results first posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Low-immersion (Mobile Device); High-immersion (Head Mounted Display)
Keywords: Virtual reality; exposure to exposure; therapist negative beliefs; exposure therapy; evidence-based practices; Simulated Exposure Trainer; virtual training program

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-immersion (mobile device) (Active Comparator)
  Interventions: Behavioral: SET-VR (computer)
- High-immersion (head-mounted display) (Experimental)
  Interventions: Behavioral: SET-VR (headset)

INTERVENTIONS:
Behavioral: SET-VR (computer) — Low-immersive version of the SET-VR program
  Arms: Low-immersion (mobile device)
Behavioral: SET-VR (headset) — High-immersive version of the SET-VR program
  Arms: High-immersion (head-mounted display)

SUMMARY:
The goal of this study is to develop a targeted virtual training program (Simulated Exposure Trainer; SET) for exposure therapy. Two platforms with differing levels of immersion (low - mobile device; high - head mounted display) will be evaluated based on their usability and engagement of an empirically-derived training target (i.e., therapist negative beliefs). Target engagement will be evaluated by applying an experimental therapeutics framework during a brief training trial.

DETAILED DESCRIPTION:
Despite the existence of numerous, well-established evidence-based practices (EBPs) for mental disorders, it has been difficult to disseminate these practices in community settings. Exposure therapy for anxiety disorders represents one of the most glaring examples of this research-to-practice gap. Just as patients are anxious about approaching their fears, therapists are often reluctant to use exposure therapy due to their own anxious beliefs that it may be dangerous and/or intolerable for patients, even after receiving specialized exposure training. Emerging training research suggests the inclusion of targeted behavioral strategies (i.e., role play, self-exposure) can reduce anxious beliefs above and beyond standard didactic training sessions. By leveraging the same behavior change principles that reduce patient anxiety (i.e., exposure), behavioral strategies can be tailored to target therapists' anxious beliefs about the treatment (i.e., conduct training as "exposure to exposure"). Unfortunately, current experiential training tasks have failed to closely replicate commonly feared clinical contexts, and as a result lack the necessary potency to potentially overcome therapist-level barriers for uptake and quality treatment delivery following training. Virtual reality (VR) has demonstrated utility as a potent and cost-effective approach for delivering exposure. We plan to investigate the application of VR as a tailored training tool (i.e., virtual "exposure to exposure" for therapists) capable of enhancing the quantity and quality of experiential learning that is lacking in current exposure training initiatives. This study will test the implementation of a VR training program on both a low-immersion (i.e., mobile device) and high-immersion (i.e., head mounted display) platform to assess which platform provides the ideal balance of immersion, usability, target engagement, and scalability. The study involves a clinical training trial to establish target engagement. Usability and target engagement information from this pilot trial will support a Phase II project aimed at building out and broadly disseminating the VR-enhanced training approach.

ELIGIBILITY:
Inclusion Criteria:

* Bachelor's level of education (or higher)
* Able to come to study site in-person for experiential training
* Has the ability to provide some sort of clinical care to patients

Exclusion Criteria:

* Found study procedures to be unacceptable during the consent process

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-07-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Anxiety Research Center at Bradley Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low-immersion (Mobile Device) | High-immersion (Head-mounted Display)
Started | 21 | 20
Completed | 21 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low-immersion (Mobile Device) | High-immersion (Head-mounted Display) | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Continuous [Mean (Full Range); unit: years] | 42 [26 to 61] | 37 [22 to 63] | 40 [22 to 63]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 2 participants did not report gender.
  Participants
    number analyzed (Participants) | 20 | 19 | 39
    Female | 17 | 17 | 34
    Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 20 | 19 | 39
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Therapist Negative Beliefs About Exposure Scale (TBES)
Description: The Therapist Negative Beliefs about Exposure Scale (TBES) assesses the extent to which therapists agree with 21 negative beliefs about exposure therapy (e.g., "most clients have difficulty tolerating the distress exposure therapy evokes"). Items are rated on a 5-point scale from 0 ("disagree strongly") to 4 ( "agree strongly"). Possible scores range from 0 to 84, with a higher score indicating more negative beliefs about exposure.
Time Frame: Before workshop starts (Baseline); immediately after 4-hour didactic portion of training (Post-didactic), immediately after remaining workshop activities (End of workshop), one month after workshop (Follow-up)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Low-immersion (Mobile Device) | High-immersion (Head-mounted Display)
Number analyzed (Participants) | 21 | 20
score on a scale
  Baseline | 28.76 (8.96) | 30.9 (10.49)
  Post-Didactic | 21.19 (10.94) | 21.2 (10.03)
  Post-Experiential | 16.33 (9.06) | 16.65 (10.50)
  Follow Up | 14.71 (10.23) | 15.95 (10.61)

2. Secondary Outcome: Exposure Self-Efficacy
Description: This is a 27-item measure of therapists' confidence in delivering exposure therapy. The first 8 items are about the therapist's ability to help patients learn skills related to exposure (e.g., "I feel confident in my ability to help my clients identify how avoidance is maintaining their fear"), and the remaining 19 items assess the therapist's confidence with implementing exposure various aspects of exposure (e.g., "I feel confident in my ability to conduct imaginal exposure"). Items are rated scale ranging from 1 ("not confident") to 5 ("very confident"). This measure has demonstrated high internal consistency and predictive validity in determining the frequency of self-reported clinical use of exposure therapy.
Time Frame: as for outcome 1
Reporting Status: Not Posted

3. Secondary Outcome: Exposure Knowledge
Description: We condensed the original 49-item Exposure Knowledge measure into 12 multiple-choice items that best fit the didactic content of the training (e.g., "Why is it important to block avoidance during exposure tasks?"). The total score is the percentage out of 100 of correct answers.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of correct answers
Arm/Group | Low-immersion (Mobile Device) | High-immersion (Head-mounted Display)
Number analyzed (Participants) | 21 | 20
percentage of correct answers
  Baseline | 42.46 (15.34) | 34.17 (15.50)
  Post-Didactic | 50.79 (18.80) | 45.83 (16.11)
  Post-Experiential | 51.98 (16.44) | 45.42 (13.91)
  Follow Up | 53.57 (18.92) | 45.83 (16.11)

ADVERSE EVENTS:
Time Frame: From enrollment through study completion (average of 2.2 months).
Description: Definitions of adverse event and/or serious adverse event used to collect adverse event information does not differ from clinicaltrials.gov definitions.
Arm/Group | Low-immersion (Mobile Device) | High-immersion (Head-mounted Display)
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 0/21 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-27): https://cdn.clinicaltrials.gov/large-docs/45/NCT06706245/Prot_SAP_000.pdf